CLINICAL TRIAL: NCT00488215
Title: A Double-Blind, Placebo-Controlled, 2-Way Cross-Over Trial in Healthy Volunteers, to Evaluate the Pharmacokinetics, Tolerability and Cardiac Safety of Oral Prucalopride at Steady State, After up-Titration to a Maximum of 20 mg.
Brief Title: A Trial in Healthy Volunteers, to Evaluate the Tolerability and Cardiac Safety of Prucalopride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: PRU-GBR-10
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2007-06

CONDITIONS: Constipation
Keywords: constipation; prucalopride; MTD; cardiovascular safety
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Prucalopride
  Interventions: Drug: prucalopride
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: prucalopride — The dose will be consecutively escalated in 2 mg steps per day, starting from 2 mg up to 20 mg once daily or until severe drug-related adverse events occur (= individual maximum tolerable dose, on decision of the subject and/or investigator).
  Other Names: Resolor
  Arms: 1
Other: Placebo — During the placebo session, the number of placebo tablets will be consecutively escalated in an identical way as described for prucalopride. This means 1 tablet more every day, up to 10 tablets.
  Arms: 2

SUMMARY:
An escalating dose of prucalopride up to a maximum of 20 mg was given once daily to 32 healthy volunteers to determine safety at the maximum tolerable dose or at 20 mg.

DETAILED DESCRIPTION:
This is a single-centre, double-blind, placebo-controlled, cross-over trial in 32 healthy volunteers with two sessions (I and II). Each session consists of a run-in day for baseline assessments, 13 treatment days and 5 additional days for assessments. Subjects will be randomized to start with either the prucalopride or placebo session.

Between the 2 sessions, there will be a washout period of 14 to 21 days, to avoid any carry-over effect.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 45 years, extremes included.
2. Subject has a normal weight as defined by a Quetelet Index range of 18 - 30 kg/m2, extremes included.
3. Informed consent form signed and dated, prior to screening.
4. Healthy on the basis of a pre-trial physical examination, medical history, anamnesis, electrocardiogram, 24 hour Holter monitoring and the results of blood biochemistry and haematology tests and a urinalysis carried out in 3 weeks preceding randomization.

Exclusion Criteria:

1. History or suspicion of alcohol, barbiturate, amphetamine or narcotic abuse.
2. Smoking more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 6 months prior to selection.
3. History of cardiac arrhythmia's, bronchospastic or cardiovascular disease (e.g. ischemic heart disease or cerebrovascular accident), diabetes mellitus, thyrotoxicosis, Parkinsonism, drug allergy.
4. Presence of prolonged QTc (Bazett) on ECG at screening (QTc > 450 msec in male subjects, QTc > 470 msec in female subjects).
5. Use of concomitant medication, except for oral contraceptives and paracetamol. All other medication must have been stopped at least 14 days before the first dose.
6. Participation in an investigational drug trial in 30 days prior to the first visit.
7. Donation of blood in the 60 days preceding the first visit.
8. Pregnancy (as confirmed by a HCG test during screening and at day 0 of each treatment session) or breast-feeding female.
9. Subjects with positive results for HIV, hepatitis B or C at screening.
10. Female subjects of childbearing potential without adequate contraceptive protection during the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2000-01; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
The exploration whether the maximum tolerable dose (MTD, defined as the highest dose not causing severe drug-related adverse events in > 50 % of the subjects) is achieved between 0 and 20 mg prucalopride. | 26 days

SECONDARY OUTCOMES:
The documentation of laboratory and cardiovascular safety (vital signs, ECG, Holter monitoring) at the MTD or at 20 mg. | 26 days

CONTACTS AND LOCATIONS:
Overall Officials: M J Boyce, M.D., Principal Investigator — Central Middlesex Hospital, London